CLINICAL TRIAL: NCT06632912
Title: A Randomized, Open-label, Non-inferiority Phase IIIb Clinical Trial to Evaluate the Immunogenicity Age/Schedule Bridging Between Adolescent Girls Aged 9-14 Years Receiving a 2-dose Regimen or Adolescent Girls Aged 9-17 Years Receiving a 3-dose Regimen of a Quadrivalent Recombinant Human Papillomavirus (HPV) Vaccine (Hansenula Polymorpha) and Women Aged 18-35 Years.
Brief Title: Phase IIIb Clinical Trial of Quadrivalent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha) for Age/Immunization Schedule Bridging
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: Chengdu Institute of Biological Products Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CNBG-CD-022-CT-4-Ⅲb
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Human Papillomavirus (HPV) Infection; HPV (Human Papillomavirus)-Associated Carcinoma
Keywords: hpv; hpv vaccine
MeSH Terms: conditions — Papillomavirus Infections; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 18-25 years old 3 doses group (Experimental)
  Interventions: Biological: 3 doses of vaccine Quadrivalent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha)
- 9-17 years old 3 doses group (Experimental)
  Interventions: Biological: 3 doses of vaccine Quadrivalent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha)
- 9-14 years old 2 doses group (Experimental)
  Interventions: Biological: 2 doses of vaccine Quadrivalent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha)
- 26-35 years old 3 doses group (Experimental)
  Interventions: Biological: 3 doses of vaccine Quadrivalent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha)

INTERVENTIONS:
Biological: 2 doses of vaccine Quadrivalent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha) — Two doses of the experimental vaccine were injected into the deltoid muscle of the upper arm according to the immunization schedule at 0 and 6 months.
  Arms: 9-14 years old 2 doses group
Biological: 3 doses of vaccine Quadrivalent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha) — Three doses of the experimental vaccine were injected into the deltoid muscle of the upper arm according to the immunization schedule at 0, 2, and 6 months.
  Arms: 18-25 years old 3 doses group; 26-35 years old 3 doses group; 9-17 years old 3 doses group

SUMMARY:
This vaccine was jointly developed by Chengdu Institute of Biological Products Co., Ltd. and National Vaccine and Serum Institute, China, is co-sponsoring this clinical trial.

This trial plans to enroll 1,800 female subjects aged 9-35 years, 450 in each of the 18-25 years old 3-dose group, 26-35 years old 3-dose group, 9-17 years old 3-dose group and 9-14 years old 2-dose group.

All subjects in the 9-14 years old 2-dose group will be injected with 2 doses of the experimental vaccine in the deltoid muscle of the upper arm according to the 0-6 month immunization schedule. Subjects in the non-immune persistence subgroup will need to complete 6 on-site visits and subjects in the immune persistence subgroup will need to complete 13 on-site visits ; All subjects in the 9-17 years old 3-dose group and the 18-35 years old 3-dose group will be injected with 3 doses of the experimental vaccine in the deltoid muscle of the upper arm according to the 0, 2, and 6 month immunization schedule. Subjects in the non-immune persistence subgroup will need to complete 9 on-site visits and subjects in the immune persistence subgroup will need to complete 16 on-site visits

ELIGIBILITY:
Inclusion Criteria:

* Females aged 9-35 years at the time of enrollment;
* Subjects aged 9-17 years at the time of enrollment and at least one legal guardian are informed and willing to participate, sign the informed consent form and can provide valid identity documents; subjects aged 18-35 years at the time of enrollment are informed and willing to participate, sign the informed consent form and can provide valid identity documents;
* Subjects are able to understand the research procedures and cooperate with the requirements of the clinical trial to participate in regular follow-up;
* Female subjects of childbearing age have a negative urine pregnancy test on the day of enrollment, are not breastfeeding and have no fertility plans within 7 months after enrollment; have taken effective contraceptive measures since the end of the last menstruation until enrollment, and agree to continue to use effective contraceptive measures within 7 months after participating in the study (effective contraceptive measures include: oral contraceptives, injections or implants, sustained-release local contraceptives, hormone patches, intrauterine devices (IUDs), sterilization, abstinence, condoms (male), diaphragms, cervical caps, etc.);
* Body temperature ≤37.0℃ (axillary temperature) on the day of enrollment.

Exclusion Criteria:

First dose exclusion criteria

* Those who have received a commercially available HPV vaccine in the past or plan to receive a commercially available HPV vaccine during the study; or have participated in other HPV vaccine clinical trials and have received the vaccine/placebo;
* Those who have a history of cervical lesions that are likely to be related to HPV infection (such as abnormal cervical cancer screening, CIN disease history); Those who have a history of hysterectomy or pelvic radiotherapy; Patients who have a history of external genital diseases that are likely to be related to HPV infection (such as vulvar intraepithelial neoplasia, vaginal intraepithelial neoplasia, and genital warts);
* Those who have a history of severe allergic reactions to any vaccine or drug (including yeast) that require medical intervention, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), etc.Or individuals with a known hypersensitivity to any of the components of the test vaccine (L-histidine, sodium chloride, aluminum hydroxide, and water for injection);
* Those who have impaired immune function or have been diagnosed with congenital or acquired immunodeficiency, human immunodeficiency virus (Human Immunodeficiency Virus). Virus, HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease or other autoimmune diseases;
* Those who have received long-term (≥14 days) immunomodulatory therapy (including immune enhancers and immunosuppressants) within 1 year prior to vaccination or within 7 months after enrollment, such as oral or injectable systemic glucocorticoid therapy (≥14 days, dose ≥2 mg/kg/day or ≥20 mg/day prednisone or equivalent prednisone dose), are permitted to use topical medications (such as ointments, eye drops, inhalers or nasal sprays), but topical medications must not exceed the dose recommended in the instructions or have any signs of systemic exposure;
* Any immunoglobulin or blood products within 3 months before vaccination or planned within 7 months after enrollment;
* Those who have received a non-live vaccine within 14 days prior to vaccination, or a live vaccine within 28 days prior to vaccination;
* Acute onset or use of antipyretic, analgesic and antiallergic drugs (such as acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) 3 days before vaccination, or acute attack of chronic diseases;
* History of convulsions (except febrile convulsions), or history or family history of epilepsy, encephalopathy, mental illness;
* Past or current severe (such as emergency treatment, surgical treatment, etc.) heart disease (such as congenital heart disease, etc.), liver and kidney disease (such as chronic hepatitis or suspected active hepatitis, nephrotic syndrome, uremia, etc.), complications of diabetes, malignant tumors, etc.;
* Elevated blood pressure measured by on-site physical examination (9-15 years old: systolic blood pressure ≥100+1.5×age (years) mmHg and/or diastolic blood pressure ≥65+age (years) mmHg; 16-26 years old: systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg);
* Participating in clinical studies of other investigational or unmarketed products (drugs, vaccines and medical devices) within 3 months before vaccination or planning to participate in the study period;
* Asplenia or functional asplenia, or splenectomy caused by any circumstances;
* Suffering from thrombocytopenia or other coagulation disorders that may be contraindications to intramuscular injection;
* Any other factors that the researcher believes make the subject unsuitable for participation in clinical trials.

Subsequent doses of vaccination should be postponed if any of the following conditions occur. Delays should ideally be made within the prescribed time window:

* Axillary temperature >37.0℃ before vaccination;
* Received any immunoglobulin or blood products within 3 months prior to vaccination;
* Received a non-live vaccine within 14 days prior to vaccination, or a live vaccine within 28 days prior to vaccination;
* Acute onset of illness or use of antipyretics, analgesics, and antihistamines (such as acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) within 3 days prior to vaccination, or an acute exacerbation of a chronic disease;
* Any other reason deemed necessary for postponement by the investigator.

If any of the following situations occur, the researcher will terminate the subsequent doses of vaccination for the subject.

* Positive urine pregnancy test before vaccination (on the day of vaccination); Note: If the subject chooses to terminate the pregnancy, at least 6 weeks after the end of the pregnancy and can submit medical evidence of termination of pregnancy (such as imaging reports or relevant medical records, etc.), the researcher can continue to vaccinate if it is considered that the subject can continue to vaccinate; if the subject chooses to continue the pregnancy, the subsequent doses of vaccination will not be administered.
* Newly discovered or newly occurring situations that meet the first dose exclusion criteria 1, 2, 3, 4, 9, 10, 13, and 14;
* After vaccination, adverse reactions related to vaccination are evaluated and considered unsuitable for continued vaccination;
* Any other reasons that the researcher assesses to terminate vaccination.

Ages: 9 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Actual)
Dates: Start 2025-11-21 (Actual); Primary Completion 2032-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titers (GMTs) of neutralizing antibodies against HPV types 6, 11, 16, and 18 among subjects who were seronegative at baseline (pre-vaccination) | 1 month after completion of the vaccination series

SECONDARY OUTCOMES:
Proportion of subjects with a ≥4-fold rise in neutralizing antibody titers against HPV types 6, 11, 16, and 18 among subjects who were seronegative at baseline (pre-vaccination) | 1 month after completion of the vaccination series
Geometric mean fold rise (GMFR) of neutralizing antibodies against HPV types 6, 11, 16, and 18 among participants who were seronegative at baseline (pre-vaccination) | 1 month after completion of the vaccination series
Geometric Mean Titers (GMTs) of neutralizing antibodies against HPV types 6, 11, 16, and 18 at 1 month after completion of the vaccination series among participants who were seropositive at baseline (pre-vaccination). | 1 month after completion of the vaccination series
Geometric mean fold rise (GMFR) of neutralizing antibodies against HPV types 6, 11, 16, and 18 among participants who were seropositive at baseline (pre-vaccination) | 1 month after completion of the vaccination series
Proportion of participants with a ≥4-fold rise in neutralizing antibody titers to HPV types 6, 11, 16, and 18 among participants who were seropositive at baseline (pre-vaccination) | 1 month after completion of the vaccination series
Geometric mean titers (GMTs) of neutralizing antibodies against HPV types 6, 11, 16, and 18 in all subjects | 1 month after completion of the vaccination series
Geometric mean fold rise (GMFR) of neutralizing antibodies against HPV types 6, 11, 16, and 18 in all subjects | 1 month after completion of the vaccination series
Proportion of subjects with a ≥4-fold rise in neutralizing antibody titers against HPV types 6, 11, 16, and 18 in all subjects | 1 month after completion of the vaccination series
Geometric mean titers (GMTs) of neutralizing antibodies against HPV types 6, 11, 16, and 18 in all subjects | 6, 12, 24, 36, 48, 60, and 72 months after completion of the vaccination series
Seropositivity rate of neutralizing antibodies against HPV types 6, 11, 16, and 18 in all subjects | 6, 12, 24, 36, 48, 60, and 72 months after completion of the vaccination series
The number of cases of AE（Adverse Event） | From the first vaccination through 1 month after completion of the vaccination series
The incidence of AEs leading to subjects withdrawing from clinical trials | From the first vaccination through 1 month after completion of the vaccination series
Distribution of severity of AE | From the first vaccination through 1 month after completion of the vaccination series
The incidence of AEs | Within 0-30 days after each vaccination (including 30 minutes, 0-7 days, and 8-30 days) and >30 days after each vaccination
Distribution of severity of AE | Within 0-30 days after each vaccination (including 30 minutes, 0-7 days, and 8-30 days) and >30 days after each vaccination
The incidence of SAE | From the first vaccination through 6 months after completion of the vaccination series
Collect information about previous pregnancies of pregnant women survey | From the first vaccination through the end of the study（Approximately 72 months）
  Such as previous pregnancy, current pregnancy mode, etc
Obtain pregnancy outcomes in pregnant subjects survey | From the first vaccination through the end of the study（Approximately 72 months）
  Collecting newborn information

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shanxian Center for Disease Control and Prevention, Heze, Shandong
  - Liaocheng Center for Disease Control and Prevention, Liaocheng, Shandong
  - Daiyue District Center for Disease Control and Prevention, Tai’an, Shandong

IPD SHARING:
Plan to Share IPD: No